CLINICAL TRIAL: NCT05015764
Title: Reprieve Cardiovascular System for the Treatment of Subjects With Acute Decompensated Heart Failure Mechanistic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reprieve Cardiovascular, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: RCV-0005
Record Dates: First submitted 2021-07-12; First posted 2021-08-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Reprieve Cardiovascular System (Experimental)
  Interventions: Device: Reprieve Cardiovascular System
- Standard of Care (Active Comparator)
  Interventions: Other: Fluid Management

INTERVENTIONS:
Other: Fluid Management — Removal of excess extracellular fluid using diuretics
  Arms: Standard of Care
Device: Reprieve Cardiovascular System — System with Fluid Management Module
  Arms: Reprieve Cardiovascular System

SUMMARY:
Reprieve Cardiovascular System for the Treatment of Subjects with Acute Decompensated Heart Failure Mechanistic Study

DETAILED DESCRIPTION:
The key objective of the trial was to provide an optimized decongestion treatment for subjects with acute decompensated heart failure and identify the critical parameters that could be incorporated into the design of the next generation of the Reprieve Cardiovascular System.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with a diagnosis of heart failure
2. Patients ≥ 18 years of age able to provide informed consent and comply with study procedures.

Exclusion Criteria:

1. Inability to place Foley catheter or IV catheter
2. Hemodynamic instability
3. Dyspnea due primarily to non-cardiac causes
4. Acute infection with evidence of systemic involvement
5. Inability to follow instructions or comply with follow-up procedures.
6. Other concomitant disease or condition that investigator deems unsuitable for the study
7. Enrollment in another interventional trial during the index hospitalization
8. Life expectancy less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Fractional Excretion of Sodium measured during therapy | End of treatment, an average of 24 hours
  Average fractional excretion of sodium across all patients measured during therapy
Device and Procedure related AEs and SAEs | Through study completion, an average of 90 days
  Rate of device and procedure related AEs and SAEs

CONTACTS AND LOCATIONS:
Locations (1):
- Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi, Georgia